CLINICAL TRIAL: NCT01238718
Title: Impact of Lidocaine on Anesthetic Depth During Rapid Sequence Induction
Brief Title: Use of Lidocaine in Rapid Sequence Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Athens (Other)
Responsible Party: University of Athens, Chryssoula Staikou, 1st department of Anesthesiology, Aretaieio Hospital, University of Athens, Greece
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: lidocaine3
Record Dates: First submitted 2010-11-08; First posted 2010-11-11 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2010-11

CONDITIONS: Hemodynamic Response
Keywords: lidocaine; anesthetic depth; hemodynamics; rapid sequence induction; BIS
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine
- normal saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine — lidocaine 1.5 mg/kg intravenously
  Arms: lidocaine
Drug: Placebo — normal saline
  Arms: normal saline

SUMMARY:
Lidocaine has been shown to blunt the cardiovascular response to endotracheal intubation. The incidence of hypertension, tachycardia and dysrhythmias due to laryngoscopy may be increased in patients that receive rapid sequence induction and intubation, where opioids are spared and intravenous anesthetic agents are not titrated step by step. Our hypothesis was that lidocaine when administered intravenously in patients who undergo rapid sequence induction may not only blunt the hemodynamic response to intubation, but may also increase the anesthetic depth (as assessed by BIS), thus further reducing the possibility of hypertension, arrhythmias and also awareness.

ELIGIBILITY:
Inclusion Criteria:

* reason for rapid sequence induction (emergency, reflux),
* ASA I-II,
* no antihypertensive drugs,
* no antiarrhythmic drugs

Exclusion Criteria :

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
BIS changes after lidocaine administration in rapid sequence induction | change from baseline in BIS values during 10 minutes

SECONDARY OUTCOMES:
change in blood pressure | change from baseline in blood pressure during 10 minutes
change in Heart rate | change from baseline in heart rate durng 10 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Aretaieio Hospital, University of Athens, Athens, Attica, Greece